CLINICAL TRIAL: NCT00560157
Title: Nutritional and Metabolic Evaluation of a Tube Feeding Immune Enhancing Diet in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCNF 0401
Record Dates: First submitted 2007-11-06; First posted 2007-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Neurological Diseases; Pneumopathy; Major Abdominal Surgery; Acute Pancreatitis
Keywords: ICU patients
MeSH Terms: conditions — Lung Diseases; Pancreatitis | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Sondalis HP
  Interventions: Dietary Supplement: Crucial (enteral tube feeding)
- II (Experimental): Crucial
  Interventions: Dietary Supplement: Crucial (enteral tube feeding)

INTERVENTIONS:
Dietary Supplement: Crucial (enteral tube feeding) — Evaluation of new enteral product, Crucial, in ICU patients

SUMMARY:
Comparison of metabolic and nutritional effects of an enteral immune enhancing diet with those of a standard polymeric one, in ICU patients

ELIGIBILITY:
Inclusion Criteria:

* 18<age<89, ASA score<4 , SAPS II score>10
* requiring the administration of an exclusive tube feeding nutrition during 7 days and beginning at the latest in the three days following the aggression
* ICU patients hospitalized for:
* neurologic affections
* pneumopathy
* major abdominal surgery or serious acute pancreatitis
* written informed consent

Exclusion Criteria:

* pregnancy or breast feeding
* immunosuppressive therapy
* radiotherapy or chemotherapy in the last six month
* uncontrolled septic choc
* auto-immune disease
* hepatic,renal or digestive insufficiency
* hyperlipidemia
* diabetes mellitus type 1
* digestive malabsorption
* life threatening situation
* treatments with growing hormone, glutamine or its metabolites or precursors such as ornithine alpha keto glutarate

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Variation of Glutamine after 90 min of enteral product administration | J5

SECONDARY OUTCOMES:
Nutritional parameters, immunologic parameters, functionality renal, Biological marker of oxidative stress | J1, J5, J8
Tolerance | Daily until J8

CONTACTS AND LOCATIONS:
Overall Officials: Luc CYNOBER, PhD, Study Chair — University PARIS V
Locations (2):
- France (2):
  - Hopital A. BECLERE, Clamart
  - Hopital Saint Antoine, Paris